CLINICAL TRIAL: NCT02918877
Title: Anesthetics to Prevent Lung Injury in Cardiac Surgery
Acronym: APLICS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Brian O'Gara, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016P000306
Record Dates: First submitted 2016-08-30; First posted 2016-09-29 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Inflammatory Lung Injury; Ischemia-Reperfusion Lung Injury; Postoperative Pulmonary Complications
Keywords: Volatile Anesthetics; Intravenous Anesthetics; Inflammatory Lung Injury; Postoperative Pulmonary Complications; Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Anesthesia (Experimental): Patients in the inhaled anesthesia arm will be given sevoflurane anesthesia maintenance for the duration of the procedure including cardiopulmonary bypass.
  Interventions: Drug: Sevoflurane
- Intravenous Anesthesia (Active Comparator): Patients in the intravenous anesthesia arm will be given total intravenous anesthesia with propofol for the duration of the procedure including cardiopulmonary bypass.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Volatile Anesthetic
  Arms: Inhaled Anesthesia
Drug: Propofol — Intravenous Anesthetic
  Other Names: Diprivan
  Arms: Intravenous Anesthesia

SUMMARY:
The purpose of this study is to investigate whether the use of inhaled anesthetics, compared to intravenous anesthetics, can affect the amount of lung inflammation and postoperative respiratory complications seen after cardiac surgery.

DETAILED DESCRIPTION:
Randomized, controlled trial involving 45 adult patients undergoing cardiac surgery with cardiopulmonary bypass. Patients will be randomized to receive either inhaled anesthesia with sevoflurane or total intravenous anesthesia (TIVA) with propofol for the maintenance phase of their cardiac anesthetic. Assessment of lung inflammation will take place using fiberoptic bronchoscopic sampling of lung fluid as well as serum collection before and after exposure to cardiopulmonary bypass, and the incidence of compositive postoperative pulmonary complications will take place in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18+)
* Undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Emergency surgery
* History of severe COPD, emphysema, or ILD
* Recent (<2wk) or current use of systemic glucocorticoids
* Prior history of pneumothorax
* Allergy/contraindication to intravenous anesthetics
* Personal or family history of malignant hyperthermia or high risk for malignant hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Gara, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Gara B, Subramaniam B, Shaefi S, Mueller A, Banner-Goodspeed V, Talmor D. Anesthetics to Prevent Lung Injury in Cardiac Surgery (APLICS): a protocol for a randomized controlled trial. Trials. 2019 May 31;20(1):312. doi: 10.1186/s13063-019-3400-x. PMID 31151474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 Enrolled
Pre-assignment Details: 49 Randomized
  * Withdrew consent (1)
  * Surgery cancelled (1)
Period: Overall Study
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Started | 24 | 25
Completed | 18 | 22
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Surgery cancelled | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Received intraoperative steroids | 1 | 0
Not completed — Unable to obtain lab samples | 1 | 0
Not completed — Unsafe to perform BAL | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (10.1) | 64.6 (10.9) | 62.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 16 | 15 | 31
  Race: Black/African American | 0 | 1 | 1
  Race: Hispanic or Latino | 2 | 3 | 5
  Race: Unknown | 0 | 3 | 3
Weight [Mean (Standard Deviation); unit: Pounds] | 207.82 (39.60) | 194.10 (42.54) | 200.96 (41.07)
Height [Mean (Standard Deviation); unit: Inches] | 69.11 (3.65) | 68.41 (3.49) | 68.76 (3.57)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.20 (4.34) | 29.61 (5.02) | 30.41 (4.68)
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 15 | 18 | 33
  Hyperlipidemia | 15 | 14 | 29
  Congestive Heart Failure | 3 | 1 | 4
  Arrhythmia | 1 | 3 | 4
  Obesity | 6 | 3 | 9
  Chronic Obstructive Pulmonary Disease/Asthma | 2 | 2 | 4
  Diabetes without Complications | 1 | 4 | 5
  Diabetes with End Organ Damage | 3 | 5 | 8
  Moderate or Severe Renal Disease | 3 | 0 | 3
  Solid (Non-Metastatic) Tumor | 3 | 2 | 5
ASA Score (American Society of Anesthesiologists) [Mean (Standard Deviation); unit: scores on a scale.] — Higher scores indicate worse preoperative comorbidity burden (on a range of 1-6).
  scores on a scale. | 3.67 (0.48) | 3.82 (0.39) | 3.75 (0.44)
ARISCAT Score [Mean (Standard Deviation); unit: scores on a scale] — Higher scores indicate worse predicted risk for postoperative pulmonary complications (range 0-123).
  scores on a scale | 50.28 (10.20) | 47.86 (8.15) | 49.07 (9.18)

OUTCOME MEASURES:

1. Primary Outcome: Bronchoalveolar Lavage (BAL) Concentration of TNF Alpha (pg/mL)
Description: Inflammatory mediator found in BAL fluid during lung inflammation
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 0.53 [0.53 to 4.99] | 0.53 [0.53 to 13.80]
  Post-Bypass | 22.06 [1.75 to 623.08] | 102.04 [2.21 to 408.05]
  Difference | 17.24 [1.22 to 536.77] | 101.51 [1.47 to 402.84]

2. Secondary Outcome: Number of Patients With Postoperative Pulmonary Complications
Description: Composite endpoint of clinically relevant pulmonary complications
Time Frame: Assessed daily, beginning on the first day after surgery, until hospital discharge or death. On average at our institution, most patients are discharged within 7 days so this is the expected time frame for follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
Participants
  Prolonged intubation (greater than 48hrs) | 0 | 3
  Failed extubation (re-intubated within 24hrs) | 0 | 1
  Reintubation (greater than 24hrs after extubation) | 0 | 2
  Pulmonary edema | 4 | 8
  Pleural effusion | 17 | 21
  Atelectasis | 16 | 19
  Infiltrate/consolidation | 6 | 6
  Pneumothorax | 1 | 5
  ARDS | 0 | 0
  Pneumonia | 0 | 1
  Brochospasm | 1 | 1
  Exacerbation of chronic lung disease | 0 | 0
  Hypoxia (PaO2/FiO2 < 300) | 16 | 15
  Respiratory acidosis (PaCO2 > 45) | 12 | 15
  Any postoperative pulmonary complication | 18 | 22

3. Secondary Outcome: BAL Concentration of IL1b (pg/mL)
Description: Inflammatory mediator found in BAL fluid during lung inflammation
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 0.42 [0.06 to 2.61] | 0.87 [0.28 to 2.54]
  Post-Bypass | 8.56 [0.21 to 64.77] | 14.37 [1.88 to 76.10]
  Difference | 8.30 [-0.67 to 59.64] | 11.00 [1.18 to 66.14]

4. Secondary Outcome: BAL Concentration of IL6 (pg/mL)
Description: Inflammatory mediator found in BAL fluid during lung inflammation
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 30.70 [6.77 to 96.60] | 31.35 [5.27 to 165.93]
  Post-Bypass | 275.19 [6.21 to 1134.33] | 297.35 [40.59 to 1277.04]
  Difference | 220.68 [-12.41 to 1046.00] | 259.32 [30.33 to 1039.58]

5. Secondary Outcome: BAL Concentration of IL8 (pg/mL)
Description: Inflammatory mediator found in BAL fluid during lung inflammation
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 2008.50 [341.25 to 16444.75] | 6528.50 [625.00 to 16332.25]
  Post-Bypass | 8019.50 [998.25 to 100438.00] | 27789.50 [4780.50 to 154087.75]
  Difference | 4701.00 [-290.25 to 77061.00] | 16230.00 [1399.25 to 123098.50]

6. Secondary Outcome: BAL Concentration of MCP1 (pg/mL)
Description: Inflammatory mediator found in BAL fluid during lung inflammation
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 509.50 [249.25 to 1415.75] | 977.50 [336.50 to 1225.75]
  Post-Bypass | 496.00 [184.25 to 2153.25] | 883.50 [651.50 to 4380.50]
  Difference | 148.00 [-265.75 to 869.75] | 479.50 [-104.25 to 1482.75]

7. Secondary Outcome: BAL Concentration of sRAGE (pg/mL)
Description: Biomarker of lung injury (RAGE - receptor for advance glycosylation end products)
Time Frame: Change from baseline and 2-4 hours after exposure to cardiopulmonary bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Number analyzed (Participants) | 18 | 22
pg/mL
  Pre-Bypass | 156.50 [44.00 to 383.00] | 164 [60.75 to 380.50]
  Post-Bypass | 597.00 [220.50 to 1195.00] | 465.00 [206.00 to 2120.50]
  Difference | 402.50 [155.25 to 1063.25] | 224.50 [-69.25 to 2088.25]

ADVERSE EVENTS:
Time Frame: During hospital length of stay ~7 days
Description: During this study, the research team did not record every adverse event. As shown in the table below (as well as the Outcome Measure 2 data), only study related events were recorded.
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 18/18 | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Anesthesia (N=18) | Intravenous Anesthesia (N=22)
Prolonged intubation (greater than 48hrs) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Failed extubation (re-intubated within 24hrs) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reintubation (greater than 24hrs after extubation) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 21 (21)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 19 (19)
Infiltrate/consolidation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Brochospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (PaO2/FiO2 < 300) (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 15 (15)
Respiratory acidosis (PaCO2 > 45) (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02918877/Prot_SAP_001.pdf